CLINICAL TRIAL: NCT06526299
Title: A Phase 2 Study of Biomarker-Modulated PSMA Theranostics
Brief Title: Low PSMA SUV Boost (LPS-Boost): Intensified 177Lu-PSMA-617 Treatment for Patients With Metastatic Castrate-Resistant Prostate Cancer With Low PSMA Expressing Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Novartis (Industry); Society of Nuclear Medicine and Molecular Imaging (SNMMI) Mars Shot Research Fund (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1124219; NCI-2024-05664 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20433 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2024-07-19; First posted 2024-07-29 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Castration-Resistant Prostate Carcinoma; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; Pluvicto; Magnetic Resonance Spectroscopy; X-Rays; Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (177Lu-PSMA-617) (Experimental): Patients receive 177Lu-PSMA-617 IV over 30 minutes on days 1, 8, 50, 57, 99 and 141. Treatment repeats every 7 days for cycles 1 and 3 and every 6 weeks for cycle 2 and subsequent cycles for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo PSMA-PET/CT during screening and SPECT/CT on study. Patients also undergo CT or MRI, bone scan, as well as blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Drug: Lutetium Lu 177 Vipivotide Tetraxetan; Procedure: Magnetic Resonance Imaging; Procedure: PSMA PET-CT Scan; Other: Questionnaire Administration; Procedure: Single Photon Emission Computed Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo SPECT/CT and CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Lutetium Lu 177 Vipivotide Tetraxetan — Given IV
  Other Names: 177Lu-labeled PSMA-617; 177Lu-PSMA-617; AAA 617; AAA-617; AAA617; Lu177-PSMA-617; Lutetium Lu 177-PSMA-617; LUTETIUM LU-177 VIPIVOTIDE TETRAXETAN; Lutetium-177-PSMA-617; Pluvicto
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: PSMA PET-CT Scan — Undergo PSMA PET/CT
  Other Names: PET-CT (PSMA); Prostate-specific Membrane Antigen PET-CT; PSMA PET-CT
Other: Questionnaire Administration — Ancillary studies
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT/CT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; Single-Photon Emission Computed; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; ST; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon

SUMMARY:
This phase II trial tests how well 177Lu-PSMA-617 works in treating patients with prostate cancer that has spread from where it first started (primary site) to other places in the body (metastatic) and that remains despite treatment (resistant). Lutetium Lu 177 (177Lu), the radioactive (tracer) component being delivered by prostate-specific membrane antigen (PSMA)-617, has physical properties that make it ideal radionuclide (imaging tests that uses a small dose tracer) for treatment of metastatic castrate-resistant prostate cancer (mCRPC). 177Lu-PSMA-617 works by binding to prostate cancer cells and inducing damage to deoxyribonucleic acid (DNA) inside prostate cancer cells. Giving 177Lu-PSMA-617 may improve treatment outcomes for patients with mCRPC.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive 177Lu-PSMA-617 intravenously (IV) over 30 minutes on days 1, 8, 50, 57, 99 and 141. Treatment repeats every 7 days for cycles 1 and 3 and every 6 weeks for cycle 2 and subsequent cycles for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo PSMA positron emission tomography/computed tomography (PET/CT) during screening and single photon emission computed tomography (SPECT)/CT on study. Patients also undergo CT or magnetic resonance imaging (MRI), bone scan, as well as blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the ability to understand and sign an approved informed consent.
* Patients must have the ability to understand and comply with all protocol requirements.
* Patients must be ≥ 18 years of age.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Patients must have a life expectancy > 6 months.
* Patients must have histological, pathological, and/or cytological confirmation of prostate cancer.
* Patients must have a positive 68Ga-PSMA PET/CT scan with no PSMA negative lesion, as determined by the Nuclear Medicine site investigator. The presence of PSMA-positive lesions was defined as 68Ga-PSMA-11 uptake greater than that of liver parenchyma in one or more metastatic lesions of any size in any organ system. PSMA negative disease defined as lymph nodes of 2.5 cm or visceral lesions or soft tissue component of a lytic bone lesion of 1.0 cm or larger with uptake less than that of liver parenchyma.
* Patients must have whole body tumor SUVmean of < 10 on 68Ga-PSMA PET/CT scan, as determined by the Nuclear Medicine site investigator. 68GaPSMA PET/CT will be analyzed using a semi-quantitative approach with MIM software (MIM Software Inc.). The workflow identified whole-body regions of interest (ROIs) with an maximum standardized uptake value (SUVmax) greater than 3 and a lesion size of at least 0.5 mm. The reviewer then manually removes any instances of physiological activity or uptake that are not related to the disease. The method of whole-body quantification will automatically calculate the whole body SUVmean.
* Patients must have prior orchiectomy and/or ongoing androgen-deprivation therapy and a castrate level of serum testosterone (< 50 ng/dL or < 1.7 nmol/L) at the most recent evaluation before enrollment.
* Patients must have received at least one androgen receptor pathway inhibitor (ARPI) (such as enzalutamide and/or abiraterone).
* Patients must have progressive mCRPC. Documented progressive mCRPC will be based on at least 1 of the following criteria:

  * Serum PSA progression defined as 2 consecutive increases in PSA over a previous reference value measured at least 1 week prior. The minimal start value is 2.0 ng/mL.
  * Soft-tissue progression defined as an increase ≥ 20% in the sum of the diameter (SOD) (short axis for nodal lesions and long axis for non-nodal lesions) of all target lesions based on the smallest SOD since treatment started or the appearance of one or more new lesions.
  * Progression of bone disease: evaluable disease or new bone lesions(s) by bone scan (2+2 Prostate Cancer Working Group 3 (PCWG3) criteria, Scher et al 2016).
* Patients must have ≥ 1 metastatic lesion that is present on baseline CT, MRI, or bone scan imaging obtained ≤ 45 days prior to beginning study therapy. Measurable disease by per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 is not required, as prostate cancer patients may not have RECIST-measurable disease but have detectable disease on bone scan.
* Patients must have recovered to ≤ grade 2 from all clinically significant toxicities related to prior therapies (i.e. prior chemotherapy, radiation, immunotherapy, etc.).
* White blood cell (WBC) count ≥ 2.5 x 10^9/L (2.5 x 10^9/L is equivalent to 2.5 x 10^3/uL and 2.5 x K/uL and 2.5 x 10^3/cumm and 2500/uL) OR absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L (1.5 x 10^9/L is equivalent to 1.5 x 10^3/uL and 1.5 x K/uL and 1.5 x 10^3/cumm and 1500/uL).
* Platelets ≥ 100 x 10^9/L (100 x 10^9/L is equivalent to 100 x 10^3/uL and 100 x K/uL and 100 x 10^3/cumm and 100,000/uL).
* Hemoglobin ≥ 9 g/dL (9 g/dL is equivalent to 90 g/L and 5.59 mmol/L).
* Total bilirubin ≤ 1.5 x the institutional upper limit of normal (ULN). For patients with known Gilbert's syndrome ≤ 3 x ULN is permitted.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 3.0 x ULN OR ≤ 5.0 x ULN for patients with liver metastases.
* Albumin > 3.0 g/dL (3.0 g/dL is equivalent to 30 g/L).
* Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min.
* HIV-infected patients who are healthy and have a low risk of AIDS-related outcomes are included in this trial. HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients who have partners of childbearing potential: Partner and/or patient must use a method of birth control with adequate barrier protection, deemed acceptable by the principal investigator during the study and for 14 weeks after last study drug administration. The patients should not donate sperm throughout the treatment period and for 14 weeks following the last treatment.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.

Exclusion Criteria:

* Previous treatment with Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223 or hemi-body irradiation within 6 months prior to treatment day 1. Previous PSMA-targeted radioligand therapy is not allowed.
* Any systemic anti-cancer therapy (e.g. chemotherapy, immunotherapy or biological therapy [including monoclonal antibodies]) within 30 days prior to treatment day 1.
* Any investigational agents within 30 days prior to treatment day 1.
* Known hypersensitivity to the components of the study therapy or its analogs.
* Other concurrent cytotoxic chemotherapy, immunotherapy, radioligand therapy, or investigational therapy.
* Transfusion within 30 days of treatment day 1.
* Patients with a history of central nervous system (CNS) metastases must have received therapy (surgery, radiotherapy, gamma knife) and be neurologically stable, asymptomatic, and not receiving corticosteroids for the purposes of maintaining neurologic integrity. Patients with epidural disease, canal disease and prior cord involvement are eligible if those areas have been treated, are stable, and not neurologically impaired.
* Symptomatic cord compression, or clinical or radiologic findings indicative of impending cord compression.
* Concurrent serious (as determined by the Principal Investigator) medical conditions, including, but not limited to, New York Heart Association class III or IV congestive heart failure, history of congenital prolonged QT syndrome, uncontrolled infection, active hepatitis B or C, or other significant co-morbid conditions that in the opinion of the investigator would impair study participation or cooperation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Prostate-specific antigen (PSA) progression-free survival (PFS) | From enrollment to PSA progression or death from any cause, assessed up to 2 years
  PSA progression is defined as a rise in PSA at > 12 weeks by more than 25% and more than 2ng/mL above the nadir (lowest PSA point). Time-to-event endpoints will be analyzed graphically and numerically using the Kaplan-Meier method and summarized in terms of median or 1-year survival point estimates with corresponding 95% confidence intervals.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days post-treatment
  AEs will be graded in severity according to the Common Terminology Criteria for Adverse Events version 5.0. Will be analyzed descriptively using summaries of counts and proportions of total and type-specific grade 3/4 AEs across cycles. The maximum toxicity grade per patient of each AE will be derived and presented in table format. The number of patients with grade 3 or higher toxicities (for each toxicity type and overall) will be provided. All AEs will be described, including clinically relevant biochemical and hematological values.
PSA50 response | Up to 30 days post-treatment
  Will be determined if an average of 70% of patients who receive the intensified regimen achieve a ≥ 50% PSA reduction in favor of the intensified regimen based on a 1-sample test of binomial proportions with 1-sided alpha = 5%. Local labs will measure PSA levels. Increases and decreases will be tracked to assess PSA responses as per Prostate Cancer Working Group 3 (PCWG3). Will be summarized as proportions with 95% confidence intervals calculated using Wilson's method and visualized using waterfall plots.
Radiographic progression-free survival | From enrollment to radiographic disease progression or death from any cause, assessed up to 2 years
  Time to radiographic progression is defined using conventional imaging or death due to any cause, whichever occurs first. Radiographic progression will be assessed per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 for soft tissue and PCWG3 for bone lesions. Will analyzed based on a 1-sample test of binomial proportions with 1-sided alpha = 5%. Time-to-event endpoints will be analyzed graphically and numerically using the Kaplan-Meier method and summarized in terms of median or 1-year survival point estimates with corresponding 95% confidence intervals.
Overall response rate (ORR) | Up to 2 years
  ORR is defined as the proportion of participants with best overall response of complete response (CR) or partial response (PR) as measured by RECIST v1.1 response in soft tissue, lymph node and visceral lesions. Will analyzed based on a 1-sample test of binomial proportions with 1-sided alpha = 5%.
Duration of response (DOR) | Up to 2 years
  DOR will also be measured in patients with a CR or PR from date of first response to the date of RECIST progression or death. Will analyzed based on a 1-sample test of binomial proportions with 1-sided alpha = 5%.
Progression-free survival (PFS) | From enrolment to first evidence of radiographic or clinical progression, or PSA PFS, assessed up to 2 years
  Clinical progression is defined as the development of signs or symptoms related to prostate cancer as assessed by the physician, initiation of other oncologic treatment or death. Will analyzed based on a 1-sample test of binomial proportions with 1-sided alpha = 5%. Time-to-event endpoints will be analyzed graphically and numerically using the Kaplan-Meier method and summarized in terms of median or 1-year survival point estimates with corresponding 95% confidence intervals.
Overall survival | From enrollment to death from any cause, assessed up to 2 years
  Will analyzed based on a 1-sample test of binomial proportions with 1-sided alpha = 5%. Time-to-event endpoints will be analyzed graphically and numerically using the Kaplan-Meier method and summarized in terms of median or 1-year survival point estimates with corresponding 95% confidence intervals.
Pain score | Up to 30 days post-treatment
  Pain will be assessed using the Brief Pain Inventory - Short Form to assess the severity of pain and the impact of pain on daily functions. Measured on Scale of 0 to 10, 0 = no pain, 10 = worst pain imaginable. Higher scores reflect more pain severity and more pain interference.
Health-related quality of life: Eastern Cooperative Oncology Group (ECOG) Performance Status scale | Up to 30 days post-treatment
  Measures one's level of functioning in terms of ability to care for oneself, daily activity, and physical ability (walking, working, etc.) with a range of 0 to 5. A score of 0 indicates performance without restriction whereas a score of 5 indicates death (a higher score indicates worse functioning).
Health-related quality of life (HRQoL): Functional Assessment of Cancer Therapy Prostate (FACT-P) | Up to 30 days post-treatment
  The FACT-P questionnaire will also be administered to assess the HRQoL of prostate cancer patients. The FACT-P is made up of 2 parts: the Functional Assessment of Cancer Therapy - General (FACT-G) questionnaire with 27 questions, and the Prostate Cancer Subscale (PCS) with an additional 12 questions. The FACT-G questionnaire measures HRQoL in four different domains: Physical well-being, Functional well-being, Emotional well-being, and Social/Family well-being. The PCS is designed specifically to measure prostate cancer-specific quality of life. Descriptive statistics will be used to summarize the original scores, as well as the change from baseline at each assessment point.
  Each item in both the FACT-G and PCS is rated on a 0 to 4 Likert-type scale, 0 being "not at all" and 4 being "very much", and then combined to produce subscale scores for each domain, as well as global quality of life score, with higher scores representing better quality of life.
Time to pain progression | From enrollment to pain progression, assessed up to 30 days post-treatment
  Will be assessed by participant responses to the Brief Pain Inventory-Short Form. Pain progression is defined as pain worsening of a 2-point or greater increase on question 3 of the inventory. Will be estimated using Kaplan-Meier method. Mean pain scores and corresponding 95% confidence intervals at each cycle will be visualized. Descriptive statistics will be used to summarize the original scores, as well as the change from baseline at each scheduled assessment time point. Additionally, changes from baseline in the scale and subscale values at the time of each assessment will be summarized. Participants with an evaluable baseline score and at least one evaluable post-baseline score during the treatment period will be included in the change from baseline analyses. The number of participants completing each questionnaire and the number of missing or incomplete assessments will be summarized for each scheduled assessment time point.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Iravani, MD FRACP, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - University of California San Francisco, San Francisco, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No